CLINICAL TRIAL: NCT06275529
Title: Evaluation of Pain and Oswestry Disability Index in Different Types of Disc Herniation According to MSU Classification in Patients Undergoing Transforaminal Epidural Steroid Injection for Radicular Low Back Pain
Brief Title: Evaluation of Transforaminal Epidural Steroid Injection in Radicular Low Back Pain According to MSU Classification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Erken, Medical Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27.12.2023.685
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Radiculopathy Lumbar; Low Back Pain; Disc Herniation; Injections, Epidural
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- MSU Classification 1A (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 1A
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 1B (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 1B
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 1C (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 1C
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 2A (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 2A
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 2B (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 2B
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 2C (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 2C
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 3A (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 3A
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 3B (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 3B
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 2AB (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 2AB
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- MSU Classification 3AB (Experimental): Transforaminal Epidural Steroid Injection, MSU classification according to MRI images 3AB
  Interventions: Procedure: Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Transforaminal Epidural Steroid Injection — Epidural injections have been used since about 1900 for the treatment of low back and lower extremity pain, with steroids added to local anesthetics in about 1950. The epidural space can be entered by 3 approaches: caudal, interlaminar, and transforaminal. Transforaminal Epidural Steroid Injections:
  After the patient is monitored in pron position and asepsis is ensured, the epidural space is entered with the appropriate needle through the transforaminal space by giving the necessary angles to the fluoroscopy. Then the location is confirmed with radiopaque agent and steroid injection is performed. The procedure takes 15-20 minutes.

SUMMARY:
Low back pain is a common disease in all ages and it effects seriously quality of life. Medical treatment,interventional methods and surgery are the treatment options. Transforaminal epidural steroid injections (TFSI) is one of the interventional method for radiculopathy with low back pain. Michigan State University(MSU) classification is a MRI based disc herniation classification. It helps to classified disc herniation in types, places and sizes.

The aim of this study to evaluate the pain and oswestry disability index in patients who have radiculopathy with low back pain, undergone TFSI according to MSU classification.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* After outpatient evaluation, a decision was made to perform transforaminal steroid injection,
* Low back pain of more than 6 on a numeric rating scale (NRS)
* Radiculopathy for more than 4 weeks and less than one year and straight leg raising <45
* Disc herniation at the L4-L5 or L5-S1 level on MRI
* Failure to respond to medical treatment for at least one month

Exclusion Criteria:

* Neurological deficit,
* Bleeding problems,
* Localized infection,
* Spinal pathologies (such as tumors),
* Fractures,
* Severe stenosis,
* Uncontrolled diabetes,
* Pregnancy,
* Red flag symptoms (such as motor and/or sphincter dysfunction)
* Patient reluctance,
* Computed tomography (CT) and MRI findings in favor of sequestrated fragments from herniated disc,
* Sphincteric disorders,
* Previous spine surgeries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change of the pain severity score | Pre-intervention, post-intervention 1th month and post-intervention 3rd month
  Pain severity is assessed by using "Numeric Rating Scale" (NRS). Patients give score of their pain between 0 (no pain) and 10 (worst possible pain).
  The change in NRS scores between the ten groups will be compared.
Change of the disability score | Pre-intervention, post-intervention 1th month and post-intervention 3rd month
  Disability conditions of the patients are assessed by using "Oswestry Disability Index" (ODI). ODI is a patient completed questionnaire which gives a percentage score of disability. The ODI is comprised of 10 items and enquires about functional limitations in various activities of daily living with the index score ranging from 1 (best) to 100 (worst).
  The change in ODI scores between the ten groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Tanyel Saraçoğlu, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No